CLINICAL TRIAL: NCT02935478
Title: A Single Center, Non-randomized Study to Evaluate the Safety and Efficacy of Left Gastric Artery Embolization in Obese Patients With Hepatocellular Carcinoma to Achieve Appropriate Weight Loss That May Allow Them to be Transplanted
Brief Title: Bariatric Embolization of Arteries in Obese Patients With HCC to Allow Salvage Liver Transplantation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB reviewing study conduct and adverse events
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Keith Pereira, MD:, MD, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27420- HCC
Record Dates: First submitted 2016-10-11; First posted 2016-10-17 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Weight Loss; Body Weight; Hepatocellular Carcinoma; HCC; Hepatitis C; Cirrhosis
Keywords: bariatric surgery; minimally invasive; Embolization; ghrelin; gastric artery embolization
MeSH Terms: conditions — Obesity; Weight Loss; Body Weight; Carcinoma, Hepatocellular; Hepatitis C; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- HCC-Left gastric artery embolization (Experimental): Embospheres Microspheres as artificial embolic agent for left gastric artery embolization
  Interventions: Device: Embospheres Microspheres

INTERVENTIONS:
Device: Embospheres Microspheres — Via a radial artery in the wrist or the femoral artery in the groin, arterial access will be obtained.Under live X-ray monitoring and using contrast, a catheter will be advanced into the artery of the stomach (left gastric artery). A CT scan will be performed on the X ray table to confirm the placement of catheter. Once this is confirmed small micro spherical particles (Embosphere Microspheres beads) will be injected though the catheter to occlude the artery and cut off blood supply to the stomach. Once the procedure is complete, in case of wrist access compression will be achieved with a band; in case of groin access a closure device will be used to plug the site of entry
  Other Names: Bariatric embolization

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common primary malignant liver tumor and has a grave prognosis. Obesity is an epidemic in the US.Patients with HCC and obesity are not candidates for liver transplantation, depriving them of the best option for cure from HCC.

Recent studies have shown that blocking blood vessels to a particular portion of the stomach (bariatric or left gastric artery embolization) can temporarily decrease levels of the appetite inducing hormone ghrelin, and result in weight loss.The purpose of this study is to determine if Left gastric artery embolization (LGAE) in patients with cirrhosis and HCC who are not transplant candidates due to morbid obesity, leads to clinically significant weight loss with eligibility for liver transplantation.

DETAILED DESCRIPTION:
Obesity:In adults, obesity is defined as a BMI of greater than 30 kg/m2. It is estimated that, by the year 2030, 38% of the world's adult population will be overweight and another 20% obese .An expert panel convened by the NIH stated that for the first time in history, the steadily improving worldwide life expectancy could level off or even decline, as the result of increasing obesity.

Liver cirrhosis with portal hypertension and HCC:

The problem: Hepatocellular carcinoma (HCC) is the most common primary malignant liver tumor seen in the setting of cirrhosis, which itself can be of varying etiology. NASH as cause for liver cirrhosis and HCC has been growing in last decade. Although Hepatitis C is currently the most common indication for liver transplant, longitudinal trends show that NASH has a trajectory to become the most common.

Current options in management: Patients who develop HCC in the context of underlying chronic liver disease complicated by portal hypertension are not candidates for resection therapy; rather, orthotopic liver transplantation (OLT) offers the best option for cure and long-term survival. Most transplant centers have strict criteria for OLT; one of the most common is a BMI < 35 kg/m2. Most NASH patients with HCC will have a high BMI. Unfortunately in presence of HCC these patients have a very limited time to lose enough weight to qualify to be listed. Lifestyle modification and medical therapies are relatively ineffective. Bariatric surgery is contraindicated in patients with portal hypertension due to significant increase in post-operative mortality, more relevant in patient listed to liver transplantation.

Thus a safe and effective minimally invasive option is needed. Based on currently available data, Left gastric artery embolization (LGAE) appears effective in inducing weight loss of about 10.5% in 3-6 months, with a high safety profile. In patients who have cirrhosis and portal hypertension with HCC and who are not transplant candidates due to morbid obesity , appropriate and timely weight loss of 10.5% in 3-6 months by performing LGAE may allow them to be listed and transplanted before their cirrhosis and tumor reaches an inoperable stage( within Milan criteria). In patients with HCC, the procedure can be performed concurrently with the procedure of Trans arterial chemoembolization which is commonly used in down staging HCC to Milan criteria.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or older.
* Willing, able and mentally competent to provide written informed consent and willing to comply with all study procedures and be available for the duration of the study
* BMI >35 kg/m2
* Adequate hematological, hepatic and renal function as follows:

  * Hematological: Platelets > 50 x 109/L, INR <1.5
  * Hepatic : Total bilirubin <3 mg/dL
  * Renal: Estimated GFR > 60ml/min.1.73m2
* Clinical, laboratory and radiographic evidence (ultrasound/ CT/MRI) of cirrhosis of any etiology with portal hypertension and concomitant HCC (treated or untreated).
* Besides a BMI >35 kg/m2, otherwise eligible for liver transplantation
* Suitable for protocol therapy as determined by the interventional radiology Investigator.

Exclusion Criteria:

* Pregnancy
* Active substance abuse
* Significant psychiatric problems, severe enough to cause suffering or a poor ability to function in life. Center for Epidemiological Studies Depression (CESD) score < 16.
* Significant alcohol consumption ( >20 g/day in women, >30 g/day in men)
* Weight > 400 lbs.
* Presence of systemic illness or other medical conditions relevant to survival .(Note that the presence of HCC will not be considered an exclusion criteria)
* Metastatic cancer
* Evidence of decompensated liver disease (uncontrolled ascites, or uncontrolled spontaneous encephalopathy)
* prior surgical weight loss procedures including gastroplasty, jejunoileal, or jejunocolic bypass, total parenteral nutrition within the past 6 months; Prior history of gastric pancreatic, hepatic, and/or splenic surgery
* Prior embolization to the stomach, spleen or liver.
* If review of available prior imaging studies (i.e. CT, MRI, or US) shows potential anatomical variations, presence of severe atheromatous disease, large arteriovenous shunting of blood.
* Abnormal Endoscopy - large sliding hiatal hernia or paraesophageal hernia, active peptic ulcer disease, active H. pylori infection
* History of abnormal Nuclear Gastric Motility examination-defined as delayed emptying of gastric contents > 90%, 60% and 10% at 1 hour, 2 hours, and 4 hours respectively.
* ASA Class 4 or 5
* Child Pugh classification C

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2017-10-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Weight | 12 months
  Total body weight loss > 10 % in 12 months

SECONDARY OUTCOMES:
Clinical parameter- Abdominal circumference | 12 months
  Improvement in abdominal circumference measured in centimeters (cm)
Clinical parameter-Blood pressure | 12 months
  Improvement in blood pressure measured in mmHg
Laboratory parameter-Ghrelin and other serum obesity hormones(Leptin, GLP-1, PYY) | 12 months
  Reduction in serum Ghrelin and other serum obesity hormones(Leptin, GLP-1, PYY) measured in pg/mL
Laboratory parameter-serum glucose | 12 months
  Reduction in serum glucose levels measured as mg/dL
Laboratory parameters- HbA1c | 12 months
  Reduction in HbA1c measures as percentage(%)
Laboratory parameters-Lipid profile | 12 months
  Improvement in lipid profile measured as mg/dL
Number of patients with clinical adverse events | 12 months
  Symptoms: pain, nausea, vomiting ;Adverse effects: Expected and unexpected
Number of patients with abnormal endoscopies | 12 months
  Photos and clinical reports analyzed for ulcers
Eligibility for liver transplant | 12 months
  Weight loss to lower BMI< 35 kg/m2 to be eligible for transplant or receive a new liver transplant.
  Proportion of patients that achieved appropriate weight reduction to be listed for transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Pereira, MD, Principal Investigator — Assistant professor of radiology-Interventional radiology; Kirubahara Vaheesan, MD, Principal Investigator — Associate professor of radiology-Interventional radiology; Alex Befeler, MD, Principal Investigator — Professor of internal medicine- Gastreoenterology; Mustafa Nazzal, MD, Principal Investigator — Assistant Professor of Surgery- abdominal transplant
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arepally A, Barnett BP, Montgomery E, Patel TH. Catheter-directed gastric artery chemical embolization for modulation of systemic ghrelin levels in a porcine model: initial experience. Radiology. 2007 Jul;244(1):138-43. doi: 10.1148/radiol.2441060790. PMID 17581899
- [Background] Arepally A, Barnett BP, Patel TH, Howland V, Boston RC, Kraitchman DL, Malayeri AA. Catheter-directed gastric artery chemical embolization suppresses systemic ghrelin levels in porcine model. Radiology. 2008 Oct;249(1):127-33. doi: 10.1148/radiol.2491071232. PMID 18796671
- [Background] Bawudun D, Xing Y, Liu WY, Huang YJ, Ren WX, Ma M, Xu XD, Teng GJ. Ghrelin suppression and fat loss after left gastric artery embolization in canine model. Cardiovasc Intervent Radiol. 2012 Dec;35(6):1460-6. doi: 10.1007/s00270-012-0362-8. Epub 2012 Feb 25. PMID 22367009
- [Background] Paxton BE, Alley CL, Crow JH, Burchette J, Weiss CR, Kraitchman DL, Arepally A, Kim CY. Histopathologic and immunohistochemical sequelae of bariatric embolization in a porcine model. J Vasc Interv Radiol. 2014 Mar;25(3):455-61. doi: 10.1016/j.jvir.2013.09.016. Epub 2014 Jan 21. PMID 24462005
- [Background] Kipshidze N, Archvadze A, Bertog S, Leon MB, Sievert H. Endovascular Bariatrics: First in Humans Study of Gastric Artery Embolization for Weight Loss. JACC Cardiovasc Interv. 2015 Oct;8(12):1641-4. doi: 10.1016/j.jcin.2015.07.016. No abstract available. PMID 26493259
- [Background] Syed MI, Morar K, Shaikh A, Craig P, Khan O, Patel S, Khabiri H. Gastric Artery Embolization Trial for the Lessening of Appetite Nonsurgically (GET LEAN): Six-Month Preliminary Data. J Vasc Interv Radiol. 2016 Oct;27(10):1502-8. doi: 10.1016/j.jvir.2016.07.010. Epub 2016 Aug 24. PMID 27567998
- [Background] Gunn AJ, Oklu R. A preliminary observation of weight loss following left gastric artery embolization in humans. J Obes. 2014;2014:185349. doi: 10.1155/2014/185349. Epub 2014 Sep 30. PMID 25349724
- [Background] Salsamendi J, Pereira K, Kang K, Fan J. Minimally invasive percutaneous endovascular therapies in the management of complications of non-alcoholic fatty liver disease (NAFLD): A case report. J Radiol Case Rep. 2015 Sep 30;9(9):36-43. doi: 10.3941/jrcr.v9i9.2557. eCollection 2015 Sep. PMID 26629307
- [Result] Olshansky SJ, Passaro DJ, Hershow RC, Layden J, Carnes BA, Brody J, Hayflick L, Butler RN, Allison DB, Ludwig DS. A potential decline in life expectancy in the United States in the 21st century. N Engl J Med. 2005 Mar 17;352(11):1138-45. doi: 10.1056/NEJMsr043743. PMID 15784668
- [Result] Chavez-Tapia NC, Tellez-Avila FI, Barrientos-Gutierrez T, Mendez-Sanchez N, Lizardi-Cervera J, Uribe M. Bariatric surgery for non-alcoholic steatohepatitis in obese patients. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD007340. doi: 10.1002/14651858.CD007340.pub2. PMID 20091629
- [Result] Hanusch-Enserer U, Brabant G, Roden M. Ghrelin concentrations in morbidly obese patients after adjustable gastric banding. N Engl J Med. 2003 May 22;348(21):2159-60. doi: 10.1056/NEJM200305223482125. No abstract available. PMID 12761382
- [Result] Mosko JD, Nguyen GC. Increased perioperative mortality following bariatric surgery among patients with cirrhosis. Clin Gastroenterol Hepatol. 2011 Oct;9(10):897-901. doi: 10.1016/j.cgh.2011.07.007. Epub 2011 Jul 23. PMID 21782772
- [Result] Lassailly G, Caiazzo R, Pattou F, Mathurin P. Bariatric surgery for curing NASH in the morbidly obese? J Hepatol. 2013 Jun;58(6):1249-51. doi: 10.1016/j.jhep.2012.12.026. Epub 2013 Jan 15. No abstract available. PMID 23333451